CLINICAL TRIAL: NCT02596048
Title: A Phase IV Multicenter Study of Iomeron®-400 Used With Multi-detector Computed Tomography Angiography (MDCTA) of the Thoraco-Abdominal Aorta, and the Carotid, Pulmonary, and Peripheral Arteries
Brief Title: A Multicenter Study of Iomeron®-400 Used With Multi-detector Computed Tomography Angiography (MDCTA)
Acronym: Iomeron®-400
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Collaborators: Bracco International B.V. (Unknown); Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IOM-122
Record Dates: First submitted 2015-10-08; First posted 2015-11-04 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Aortic Disorders; Carotid Disease; Pulmonary Disease; Peripheral Artery Disease
MeSH Terms: conditions — Aortic Diseases; Lung Diseases; Peripheral Arterial Disease | interventions — iomeprol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iomeron (Other): Patients will undergo a injection of Iomeron if they are scheduled to undergo an elective thoraco-abdominal aorta, carotid, pulmonary or peripheral MDCTA examination
  Interventions: Other: Iomeron

INTERVENTIONS:
Other: Iomeron — Iomeron or Imeron which is a iomeprol injection, hereafter referred to as iomeprol is an injectable solution of iomeprol, a non-ionic hydrosoluble iodinated compound used as a medical imaging contrast agent for radiological examinations.
  Other Names: iomeprol injection; Imeron

SUMMARY:
This is a Phase IV multicenter, open-label study and is being implemented in order to assess diagnostic image quality of MDCTA in subjects undergoing computed tomography angiography (CTA) of the thoraco-abdominal aorta, and the carotid, pulmonary and peripheral arteries with IOMERON.

DETAILED DESCRIPTION:
This is a Phase IV multicenter, open-label study and is being implemented in order to assess diagnostic image quality of MDCTA in subjects undergoing computed tomography angiography (CTA) of the thoraco-abdominal aorta, and the carotid, pulmonary and peripheral arteries with IOMERON. The hypothesis is that IOMERON used at a high concentration will provide good diagnostic image quality. The Investigators will also function as readers and evaluate the images on-site. Efficacy analysis will be based on the on-site evaluations.

Imaging conditions will be representative of those used in routine clinical practice. The study will be conducted at approximately 10-20 sites in China. Each site may enroll approximately 40 subjects in this study. Approximately 400 subjects will be enrolled in order to obtain 360 evaluable subjects who undergo elective MDCTA of the thoraco-abdominal aorta, or carotid, pulmonary or peripheral arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Provides written Informed Consent and is willing to comply with protocol requirements
2. Is at least 18 years of age.
3. Is scheduled to undergo an elective thoraco-abdominal aorta, carotid, pulmonary or peripheral MDCTA examination.

Exclusion Criteria:

1. Is a pregnant or lactating female. Exclude the possibility of pregnancy:

   by testing on site at the institution (serum or urine βHCG) within 24 hours prior to the start of investigational product administration, by surgical history (e.g., tubal ligation or hysterectomy),post-menopausal with a minimum 1 year without menses;
2. Has any known allergy to one or more of the ingredients of IOMERON or a history of hypersensitivity to iodinated contrast agents;
3. Has moderate to severe renal impairment;
4. Has received an investigational compound and/or medical device within 30 days before admission into this study;
5. Has been enrolled previously to this study
6. Has any medical condition or other circumstances which would significantly decrease the chances of obtaining reliable data, achieving study objectives, or completing the study and/or post-dose follow-up examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2015-12; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with an 3 point scoring system used for assessing diagnostic image quality | 2 hours
  0 = Insufficient: Impaired image quality precludes adequate diagnostic assessment of vascular abnormalities (stenosis, embolism, dissection, etc.) because of severe noise, or severe artifacts, or insufficient contrast enhancement.
  1. = Adequate: Image quality is sufficient for adequate diagnostic assessment of vascular abnormalities (stenosis, embolism, dissection etc.), even in presence of minimal noise, or minimal artifacts and sufficient contrast enhancement.
  2. = Good: Image quality allows adequate, complete and rapid diagnostic assessment of vascular abnormalities (stenosis, embolism, dissection etc.) with absent or very minimal noise, or absent or very minimal artifacts, and optimal contrast enhancement.
Number of participants with an 3 point scoring system used for visual assessment of contrast enhancement and delineation of vascular structures/abnormalities | 2 hours
  0 = Insufficient: Generally poor enhancement and delineation of major vascular structures/abnormalities (e.g. major endoleaks, aneurysms, bleeding, etc.).
  1. = Adequate: Sufficient enhancement and delineation of vascular structures/abnormalities (e.g. small bleeding, endoleaks, etc).
  2. = Good: Optimal enhancement and complete delineation of vascular structures/abnormalities (e.g. small bleeding, endoleaks, etc).

SECONDARY OUTCOMES:
Comparing number of participants undergoing x-ray angiography as the truth standard with the diagnostic performance of MDCTA diagnosis using a two point scoring system | 2 hours
  0 = Inadequate: Relevant aspects of MDCTA diagnosis do not match with the truth standard
  1 = Adequate: Relevant aspects of the MDCTA diagnosis match with the truth standard

CONTACTS AND LOCATIONS:
Overall Officials: Martin Krix, MD, MSc, Study Director — Bracco Imaging Deutschland
Locations (5):
- China (5):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Wuhan Union Hospital, Wuhan, Hubei
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Affiliated Hospital of Xi'an Jiaotong University, Shanxi Province, Shanxi
  - The First Teaching Hospital of Xinjiang Medical University, Ürümqi, Xinjiang

REFERENCES:
- [Background] Fleischmann D. High-concentration contrast media in MDCT angiography: principles and rationale. Eur Radiol. 2003 Nov;13 Suppl 3:N39-43. doi: 10.1007/s00330-003-0005-1. No abstract available. PMID 15015879
- [Background] Bae KT. Intravenous contrast medium administration and scan timing at CT: considerations and approaches. Radiology. 2010 Jul;256(1):32-61. doi: 10.1148/radiol.10090908. PMID 20574084